CLINICAL TRIAL: NCT02638766
Title: Phase II, Single Arm, Non-randomized and Multicenter Clinical Trial of Regorafenib as a Single Agent in the First-line Setting for Patients With Metastatic and/or Unresectable KIT/PDGFR Wild Type GIST
Brief Title: Single Agent Regorafenib in First-line for Metastatic/Unresectable KIT/PDGFR Wild Type GIST
Acronym: REGISTRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGISTRI (GEIS 40)
Record Dates: First submitted 2015-11-11; First posted 2015-12-23 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: metastatic; unresectable; KIT/PDGFR wild type GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unique arm (Other): Regorafenib 160mg once a day, frequency: 3 weeks on/1 week off in cycles of 28 days
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib — Treatment with regorafenib 160mg once a day, 3 weeks on / 1 week off in cycles of 28 days
  Other Names: Stivarga

SUMMARY:
Evaluate the treatment with regorafenib in patients with metastatic and/or unresectable KIT/PDGFR wild type GIST in the first line setting.

DETAILED DESCRIPTION:
The SDH complex is involved in mitochondrial Krebs cycle and defects in the succinate dehydrogenase (SDH) complex have identified, as previously mentioned, in KIT/PDGFR WT. This complex, SDH, has 4 subunits (A-D) and SDH-A or SDH-B are involved in oxidization succinate to fumarate. Therefore, loss of function owing to mutational inactivation leads to the cytoplasmic accumulation of succinate which downregulates prolyl hydroxylase. This enzyme has a negative regulator role of hypoxia-inducible factor 1α (HIF1α) since promotes its proteasomal degradation. Increased levels of HIF1α can enter the nucleus and activate the transcription of vascular endothelial growth factor (VEGFR)24. In fact, the VEGFR expression is higher in KIT/PDGFR WT than in KIT mutant GISTs25.

Approximately 50% of KIT/PDGFR WT show high expression of insulin-like growth factor 1 receptor (IGFR1). This expression may correlate also with the loss of SDH due to IGF autocrine loop26. IGFR signals through both MAPK and PI3K-AKT pathways. As previously mentioned, Regorafenib is able to block MAPK signaling pathway at different levels. Interestingly, early interstitial Cajal cell (ICC) progenitors have a phenotype of KITlowCD44+CD34+IGFR+ while committed lineage of progenitors have KIThighCD44+CD34-IGFR-. Unlike mature or more committed lineage of ICCs, the KITlowCD44+CD34+IGFR+ display resistance to Imatinib in spite of kit signaling pathway activation. Thus Regorafenib could gain advantage over Imatinib for treating KIT/PDGFR WT27,28.

On the other hand, other subsets within of KIT/PDGFR WT as B-RAF mutants or NF1-associated GIST could also be sensitive to Regorafenib. In this later subset, protein expression of phospho-MAPK was seen in 92% of cases in a series of 25 patients29.

Theoretically Regorafenib could also act blocking STAT3, which is activated by RET proto-oncogen, through RET inhibition. STAT3 is implicated as downstream pathway signal in GIST30.

Taken together, the previous data suggests Regorafenib could play a relevant role as upfront treatment of metastatic or unresectable locally advanced KIT/PDGFR WT GIST.

Subjects will receive 160mg (4 tablets) of regorafenib once a day every day for 3 weeks of every 4 week cycle (i.e., 3 weeks on, 1 week off). The study drug will be orally administered.

Doses of study drug may be delayed or reduced in case of clinically significant hematologic and other toxicities. Toxicities will be graded using the CTCAE v 4.03. The modifications of regorafenib are detailed in the protocol for general event, Hand Foot Skin Reaction, Hypertension and drug-related liver function test abnormalities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up.

   Informed Consent must be obtained prior to start of the screening process. Procedures conducted as part of the patient´s routine clinical management (e.g. blood count, imaging tests, etc.) and obtained prior to signature of informed consent may be used for screening or baseline purposes as long as these procedures are conducted as specified in the protocol.
2. Male or female subjects ≥18 years of age
3. Histologically confirmed GIST KIT/PDGFR wild-type, unresectable or metastatic GIST (confirmed by central laboratory). Paraffin-embedded tumor block must be provided by all subjects during screening period.
4. Screening of mutations done in exon 11, 9, 13 and 17 in KIT gene and in 12 and 18 exons of PDGFR gene
5. Subjects must have at least one measurable lesion according to RECIST v1.1 criteria. A lesion in a previously irradiated area is eligible to be considered as measurable disease as long as there is objective evidence of progression of the lesion prior to study enrolment.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
7. Adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:

   * Total Bilirubin ≤ 1.5 x the upper normal limit (UNL). Documented Gilbert Syndrome is allowed if total bilirubin is mildly elevated (≤6mg/dl).
   * Alanine Aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x UNL (≤5xUNL for subjects with liver involvement of GIST)
   * Lipase ≤1.5 x UNL
   * Serum Creatinine ≤ 1.5 x UNL
   * Glomerular filtration rate (GFR) ≥ 30ml/mn/1.73 m2 according to the Modified Diet in Renal Disease (MDRD) abbreviated formula.
   * International Normalized Ratio (INR) ≤1.5xUNL and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤1.5xUNL. Subjects who are being treated with an anti-coagulant, such as warfarin or heparin, will be allowed to participate provided that no prior evidence of an underlying abnormality in these parameters exists. Close monitoring of at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standards of care.
   * Platelet count ≥100000mm3, hemoglobin (Hb) ≥ 9.0 g/dl, absolute neutrophil count (ANC) ≥1500/mm3. Blood transfusions to meet the inclusion criteria will not be allowed.
   * Alkaline phosphatase limit ≤ 2.5 x UNL (≤ 5x UNL for subjects with disease involving the liver)
8. Women of childbearing potential and men must agree to use adequate contraception from the moment of signing the Informed Consent Form until at least 3 months after the last study drug administration. The investigator or a designated associate is requested to advise the subject on how to achieve an adequate birth control. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care.
9. Women of childbearing potential must have a blood or urine pregnancy test performed a maximum of 7 days before start of study treatment, and a negative result must be documented before start of study treatment.

Exclusion Criteria:

1. Prior systemic treatment for GIST BESIDES IMATINIB. Patients that have relapsed after receiving imatinib during adjuvant setting and patients who are on treatment or have been treated with Imatinib as first line of advanced KIT/PDGFRa wild type GIST are eligible.
2. Cancer other than GIST within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, and superficial bladder tumors (Ta (Non Invasive tumor), and Tis (Carcinoma In situ)).
3. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before the start of study medication.
4. Congestive Heart Failure New York Heart Association (NYHA) ≥ class 2.
5. Unstable angina (angina symptoms at rest, new-onset angina, ie, within the lasts 3 months prior to entering study) or myocardial infarction (MI) within the past 6 months before the start of study medication.
6. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
7. Uncontrolled hypertension (Systolic blood pressure > 140 mmHg or diastolic pressure > 90mmHg despite optimal medical management).
8. Subjects with pheochromocytoma.
9. Arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), or pulmonary embolism within 6 months from start of study treatment.
10. Venous thrombotic events such as deep vein thrombosis within the 3 months before the start of study treatment.
11. Ongoing infection > grade 2 National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03
12. Known history of human immunodeficiency virus (HIV) infection.
13. Subjects with seizure disorder requiring medication
14. Symptomatic metastasis in brain or meningeal tumors.
15. History of organ allograft.
16. Subjects with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ NCI-CTCAE version 4.03 grade 3 or higher within 4 weeks prior to start of study treatment.
17. Non-healing wound, ulcer, or bone fracture.
18. Renal failure requiring hemo- or peritoneal dialysis.
19. Dehydration NCI-CTCAE version 4.03 grade ≥ 1
20. Substance abuse or medical, psychological, or social conditions that may interfere with the subject´s participation in the study or evaluation of the study results.
21. Known hypersensitivity to the study drug, study drug class, or excipients in the formulation.
22. Any illness or medical conditions that are unstable or could jeopardize the safety of the subject and his/her compliance in the study
23. Interstitial lung disease with ongoing signs and symptoms at the time of screening.
24. Subjects unable to swallow oral medication
25. Persistent proteinuria of NCI-CTCAE version 4.03 grade 3 or higher (>3.5g/24hrs), measured by urine protein creatinine ratio on a random urine sample)
26. Any malabsorption condition.
27. Left Ventricular Ejection Fraction (LVEF) < 50% or below the LLN for the institution (whichever is higher).
28. Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE version 4.03 grade 2 dyspnea)

NOTE: It is not necessary to demonstrate disease progression or imatinib intolerance to offer the study entrance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11; Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate | every 8 weeks during 36 months
  the sum of complete responses (CR) + partial responses (PR) + stable disease (SD).

SECONDARY OUTCOMES:
Progression free survival | every 8 weeks during 36 months
  Number of months without progression
Overall survival | Every 8 weeks during 36 months
  Number of months alive
Responses determined by CHOI | every 8 weeks during 36 months
  Measure tumor size
Correlation with translational research | After 36 months of recruitment
  Relation between the clinical data obtained and the data obtained from translational research
Safety (adverse events following CTCAE v4.03) | Every 28 days until 30 days after last dose
  Evaluation of adverse events following CTCAE v4.03
Early metabolic response by PET scan | After 1 month of starting treatment
  Evaluation of metabolic response to treatment
Quality of life by EORCT QLQ C30 questionnaire | Day 1 of each cycle. Pre-treatment administration
  EORCT QLQ C30 questionnaires
Quality of life by EQ-ED-5L questionnaire | Day 1 of each cycle. Pre-treatment administration
  EQ-ED-5L questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martín-Broto, MD, Study Chair — GEIS (GRUPO ESPAÑOL DE INVESTIGACION EN SARCOMAS; Virginia Martínez-Marín, MD, Study Director — GEIS (GRUPO ESPAÑOL DE INVESTIGACION EN SARCOMAS
Locations (17):
- France (3):
  - Institute Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Gustave Roussy, Villejuif
- Italy (4):
  - Fondazione IRCCS Istituto Dei Tumori di Milano, Milan
  - Fondazione G Pascale Napoli, Napoli
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Istituto di Candiolo - IRCSS, Torino
- Spain (10):
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital de Cruces, Barakaldo
  - Hospital Universitario Vall d´hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen de la Macarena, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin-Broto J, Valverde C, Hindi N, Vincenzi B, Martinez-Trufero J, Grignani G, Italiano A, Lavernia J, Vallejo A, Tos PD, Le Loarer F, Gonzalez-Campora R, Ramos R, Hernandez-Jover D, Gutierrez A, Serrano C, Monteagudo M, Leton R, Robledo M, Moura DS, Martin-Ruiz M, Lopez-Guerrero JA, Cruz J, Fernandez-Serra A, Blay JY, Fumagalli E, Martinez-Marin V. REGISTRI: Regorafenib in first-line of KIT/PDGFRA wild type metastatic GIST: a collaborative Spanish (GEIS), Italian (ISG) and French Sarcoma Group (FSG) phase II trial. Mol Cancer. 2023 Aug 9;22(1):127. doi: 10.1186/s12943-023-01832-9. PMID 37559050